CLINICAL TRIAL: NCT02261207
Title: Phase II Study on Axitinib in Advanced VEGFR and/or PDGFR Solitary Fibrous Tumor
Brief Title: Phase II Study on Axitinib in Advanced Solitary Fibrous Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SFT-AX2014; 2013-005596-40 (EudraCT Number)
Record Dates: First submitted 2014-01-30; First posted 2014-10-10 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Solitary Fibrous Tumor
MeSH Terms: conditions — Solitary Fibrous Tumors | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Axitinib (Experimental): Axitinib will be administered at the dose of 5mg twice a day, continuously. Treatment will be continued till evidence of progression, or toxicities or patient withdrawal.
  Interventions: Drug: Axitinib

INTERVENTIONS:
Drug: Axitinib — Axitinib will be administered at the dose of 5mg twice a day, continuously. Treatment will be continued till evidence of progression, or toxicities or patient withdrawal.
  Other Names: Inlyta

SUMMARY:
This is an investigator initiated, open label, prospective, non-randomized, phase II trial aimed at evaluating the activity of Axitinib in progressive VEGFR2 and/or PDGFRB positive advanced Solitary Fibrous Tumor (SFT) patients. Patients with a documented and centrally reviewed pathologic and radiologic diagnosis of progressive VEGFR2 and/or PDGFRB positive advanced SFT may enter in the study. Axitinib will be administered at the dose of 5mg twice a day, continuously. Treatment will be continued till evidence of progression, or toxicities or patient withdrawal.

DETAILED DESCRIPTION:
This is an investigator initiated, open label, prospective, non-randomized, phase II trial aimed at evaluating the activity of Axitinib in progressive VEGFR2 and/or PDGFRB positive advanced Solitary Fibrous Tumor (SFT) patients. Patients with a documented and centrally reviewed pathologic and radiologic diagnosis of progressive VEGFR2 and/or PDGFRB positive advanced SFT may enter in the study. Axitinib will be administered at the dose of 5mg twice a day, continuously. Treatment will be continued till evidence of progression, or toxicities or patient withdrawal.

The activity of Axitinib will be evaluated in terms of overall response rate according to Choi Criteria as defined for GIST patients treated with Imatinib, extended even to MRI.

Secondary objectives of the study will be: response rate by RECIST, progression free survival, overall survival, clinical benefit (RECIST Complete Response + Partial Response + Stable Disease >6 months). Whenever possible a post-treatment biopsy will be performed to assess Axitinib targets status after treatment and to correlate their status to the response.

Tumor assessment with CT scan and/or MRI will be performed within 4 weeks prior to first dose of Axitinib and after 4 weeks from starting treatment, then every 2 months until progression or toxicity.

As per protocol the experimental treatment can be administered in front or further line.

The study will be considered positive if 30% of response rate by Choi criteria is observed. To this end a maximum of 16 evaluable patients will be enrolled in two years.

In case of positive study the trial will be re-open to confirm the result in a larger number of patients.

.

ELIGIBILITY:
Inclusion Criteria:

* Pat centrally confirmed diagnosis of solitary fibrous tumor
* Expression of PDGFRB and/or VEGFR2 by immunohistochemistry on formalin fixed-paraffin embedded (FFPE) material as minimal requirement. Activation of PDGFRB and/or VEGFR2 by real time C reactive protein of PDGFB and VEGFA on FFPE material (if in sufficient quantity) or by biochemistry on frozen material (if available)
* Locally advanced disease (i.e. surgical resection of local disease unfeasible radically, or unaccepted by the patient, or amenable to become less demolitive, or feasible, or easier, after cytoreduction) and/or metastatic disease
* Measurable disease
* Centrally confirmed evidence of progression by RECIST during the 6 months before study entry
* 1st-line vs 3-rd-line
* Eastern Cooperative Oncology Group (ECOG) Performance Status = 0, 1, 2
* Adequate bone marrow function, defined as the following: absolute neutrophil count (ANC) >1.5 x 109/L, platelets >100 x 109/L, Hb >9 g/dL. Blood transfusions are allowed to reach the baseline requested Hb level
* Adequate organ function, defined as the following: total bilirubin within normal institutional limits (but in case of Gilbert's syndrome), aspartate aminotransferase (AST) and Serum Glutamic Pyruvic Transaminase (ALT) <2.5 x upper normal limit (UNL), creatinine <1.5 x upper normal limit (UNL), within normal institutional limits or creatinine clearance ≥60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Cardiac ejection fraction ≥50% as measured by echocardiogram
* Age > 18 yrs
* Female patients of child-bearing potential must have negative pregnancy test within 7 days before initiation of study drug dosing. Post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients of reproductive potential must agree to employ an effective method of birth control throughout the study and for up to 3 months following discontinuation of study drug
* No history of arterial and/or venous thromboembolic event within the previous 12 months
* Written, voluntary informed consent

Exclusion Criteria:

* Other primary malignancy with <5 years clinically assessed disease-free interval, except basal cell skin cancer, cervical carcinoma in situ, or other neoplasms judged to entail a low risk of relapse
* Previous treatment with any other investigational or not investigational agents and or radiation therapy within 28 days of first day of study drug dosing, or patients who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Major surgery within 2 weeks prior to study entry
* Previous radiotherapy to ≥25 % of the bone marrow
* Concomitant other investigational agents or concurrent anticancer therapy. In addition, all herbal (alternative) medicines are excluded
* Grade III/IV cardiac problems as defined by the New York Heart Association Criteria (i.e., history of uncontrolled or symptomatic angina, history of arrhythmias requiring medications, or clinically significant, with the exception of asymptomatic atrial fibrillation requiring anticoagulation, myocardial infarction < 6 months from study entry, uncontrolled or symptomatic congestive heart failure, ejection fraction below the institutional normal limit)
* Known chronic liver disease (i.e., chronic active hepatitis, and cirrhosis with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
* Known diagnosis of human immunodeficiency virus (HIV) infection
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Axitinib
* Expected non-compliance to medical regimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-11; Primary Completion 2017-10 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Response rate by Choi criteria | 4 years
  response rate, according to Choi Criteria

SECONDARY OUTCOMES:
Response rate by RECIST criteria | 4 years
  response rate according to RECIST

OTHER OUTCOMES:
Overall survival | 4 years
  Evaluation of overall survival
Progression Free Survival | 4 years
  Evaluation of Progression Free Survival
Clinical Benefit | 4 years
  Evaluation of clinical benefit according to response rate, overall survival, progression free survival
Post-treatment Axitinib target status assessment | 4 years
Safety essessment | 4 years
  assessment of the safety profile of Axitinib in agreement with the incidence of related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Stacchiotti, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Naazionale dei Tumori, Milan, MI, Italy